CLINICAL TRIAL: NCT03214835
Title: CDx Biopsies for Detection of Laryngopharyngeal Reflux and Laryngeal Lesions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant.
Sponsor: CDx Diagnostics (Industry)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CDx Laryngeal and LPR Study
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Laryngeal Disease; Laryngeal Tumor; Laryngopharyngeal Reflux
Keywords: Larynx; reflux; LPR; tumor; lesion
MeSH Terms: conditions — Laryngeal Diseases; Laryngopharyngeal Reflux; Gastroesophageal Reflux; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brush biopsy for laryngeal lesion (Experimental): Brush biopsy of the larynx - in addition to the standard biopsy
  Interventions: Device: Endo CDx Brush biopsy
- Brush biopsy for LPR (Experimental): Brush biopsy of the larynx at the post cricoid region - in addition to the standard examination for LPR (PH monitoring double probe)
  Interventions: Device: Endo CDx Brush biopsy

INTERVENTIONS:
Device: Endo CDx Brush biopsy — In patients with laryngeal lesion the brush biopsy will be taken with the standard cup biopsy - either in the clinic or in the OR. In LPR patients brush biopsy will be taken in the clinic.

SUMMARY:
The study will take place at Rambam medical center, department of Otolaryngology Head and Neck Surgery, for two years. Patients suspected of LPR or laryngeal l tumor and are candidate for laryngeal or hypopharyngeal biopsies will be recruited.

DETAILED DESCRIPTION:
First- all patients visiting our clinic with laryngeal complaints suspicious for either LPR or laryngeal tumor will fill the RSI questionnaire. Then fiberoptic examination will be performed by a laryngologist that will complete the RFS score.

Patients with suspicious lesions will be referred for TFL standard biopsy and CDx brush biopsy in order to determine whether the lesions are malignant or benign. The pathologic diagnosis of invasive carcinoma from a TFL biopsy is considered equivalent to the pathology results from a direct laryngoscopy biopsy. All patients with benign pathology or carcinoma in-situ (CIS) on TFL biopsy will be referred for subsequent direct laryngoscopy (DL) for definitive diagnosis. At the time of the DL biopsy will include also another CDx brush smear. Patients with benign-appearing lesions will be taken for lesion removal and biopsy.Before removal of the lesion a CDx brush smear will be collected.

All the participants suspected of LPR will have: PHmetry with Manometry andCDx brush biopsy.All relevant demographic and clinical data will be retrieved for analysis.

CDx biopsies will be an addition to the routine management of the patients in the diagnosis and follow-up of laryngeal lesions and LPR and will not replace the standard regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* patients suspected to suffer from LPR
* Patients with laryngeal/hypopharyngeal lesions.

Exclusion Criteria:

* Patient refusal
* Patients with anatomical variants which precludes biopsy taking.
* Patients with allergy to lidocain-based local anesthesia agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of EndoCDx brush | 3 months
  Efficacy of EndoCDx brush biopsy as a diagnostic tool for laryngeal lesions compared to cup forceps biopsy and a diagnostic tool for LPR compared to double probe PH monitoring

SECONDARY OUTCOMES:
Assessment of pain | 6 months
  Assessment of pain during EndoCDx brush biopsy under local anesthesia by Visual Analog Score for pain

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Cohen, MD, Principal Investigator — Rambam Health Care Campus